CLINICAL TRIAL: NCT06672094
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of NeuroQ on Cognitive Function in Healthy Adults with Self-reported Memory Problems.
Brief Title: A Study to Investigate the Safety and Efficacy of NeuroQ on Cognitive Function in Health Adults with Self-Reported Memory Problems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LifeSeasons Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23LSCNF01
Record Dates: First submitted 2024-10-24; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Self-reported Memory Problems

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeuroQ (Experimental): Participants will be instructed to take two (2) capsules of NeuroQ every morning with or without food starting on Day 1. Clinic staff will instruct participants to save all unused and open packages and return them to KGK Science Inc. for a determination of compliance. If a dose is missed participants are instructed to re-start their regular dosing the next day and document the missed dose in their study diary. Participants will be advised not to exceed two capsules daily.
  Interventions: Dietary Supplement: NeuroQ
- Placebo (Placebo Comparator): Participants will be instructed to take two (2) capsules of placebo every morning with or without food starting on Day 1. Clinic staff will instruct participants to save all unused and open packages and return them to KGK Science Inc. for a determination of compliance. If a dose is missed participants are instructed to re-start their regular dosing the next day and document the missed dose in their study diary. Participants will be advised not to exceed two capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NeuroQ — Two (2) capsules of NeuroQ taken once a day for 60 days.
  Arms: NeuroQ
Other: Placebo — Two (2) capsules of placebo taken once a day for 60 days.
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the safety and efficacy of NeuroQ on cognitive function in a North American population of healthy adults with self-reported memory problems compared to placebo. The difference in change in cognitive function as assessed by the CNS Vital Signs (CNS VS) Neurocognitive Index (NCI) score between NeuroQ and placebo will be measured from baseline at Day 60. Additionally, the safety and tolerability of NeuroQ, as compared to placebo, will be measured by the occurrence of and/or changes in treatment-emergent adverse events (AEs). Participants will take two capsules containing NeuroQ or placebo once a day for 60 days, have 4 in-person clinic visits, and keep a diary of their symptoms and number of missed doses.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 40-79 years of age, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active
3. Individuals with self-reported memory problems as assessed by a combined score of ≥6 on Everyday Memory Questionnaire questions 1, 2 and 18 at screening
4. Absence of dementia or other significant cognitive impairment as assessed by Mini Mental State Examination-2 Standard Version (MMSE-2) score ≥24 at screening
5. Agrees to avoid high sources of caffeine (e.g., supplements, tea, coffee, energy drinks), NSAIDs, and alcohol consumption for 24 hours prior to in-clinic visits
6. Agrees to avoid first generation anti-allergy medication for 48 hours prior to in-clinic visits
7. Agrees to avoid moderate-vigorous exercise 12 hours prior to in-clinic visits
8. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
9. Willing and able to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history, laboratory results, and vital signs, as assessed by the QI

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product or placebo ingredients
3. Self-reported confirmation of any significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
4. Self-reported color blindness/weakness as assessed by the QI
5. Individuals who consume high caffeine daily or are addicted to caffeine at screening as assessed by the QI
6. Individuals with >2 chronic diseases and/or acute disease as assessed by the QI
7. Individuals with amyloidosis and/or cystinuria
8. Current employment that calls for overnight shiftwork as assessed by the QI
9. Travel across two or more time zones two weeks prior to any study visit
10. Unstable metabolic disease or chronic diseases as assessed by the QI
11. Current or history of significant diseases of the gastrointestinal tract or conditions that result in malabsorption, as assessed by the QI
12. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3.1)
13. Type I diabetes
14. Type II diabetes if on insulin treatment. Type II diabetics on stable medication for at least three months and an HbA1c of <8.0% may be included after assessment by the QI on a case-by-case basis
15. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
16. History of or current diagnosis with kidney, gallbladder (e.g., gallstones, bile duct obstruction), and/or liver diseases (e.g., reduced bile salts, SIBO) as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
17. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
18. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
19. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
20. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
21. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
22. Self-reported confirmation of blood/bleeding disorders as assessed by QI
23. Use of medical cannabinoid products
24. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
25. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
26. Alcohol intake average of >2 standard drinks per day as assessed by the QI
27. Alcohol or drug abuse within the last 12 months
28. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Sections 7.3.1 and 7.3.2)
29. Clinically significant abnormal laboratory results at screening as assessed by the QI
30. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
31. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
32. Individuals who are cognitively impaired and/or unable to give informed consent
33. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
The difference in change in cognitive function between NeuroQ and placebo. | baseline (day 0) and 60 days
  The difference in change in cognitive function as assessed by the CNS Vital Signs (CNS VS) Neurocognitive Index (NCI) score between NeuroQ and placebo from baseline at Day 60

SECONDARY OUTCOMES:
The difference in change in cognitive function between NeuroQ and placebo in NCI score | baseline (day 0) and 7 days
  The difference in change in cognitive function as assessed by the CNS VS between NeuroQ and placebo in NCI score from baseline at Day 7
The difference in change in cognitive function between NeuroQ and placebo in individual domain scores | baseline (day 0) and 7 days
  The difference in change in cognitive function as assessed by the CNS VS between NeuroQ and placebo in individual domain scores from baseline at Day 7
The difference in change in cognitive function between NeuroQ and placebo in individual domain scores | baseline (day 0) and 60 days
  The difference in change in cognitive function as assessed by the CNS VS between NeuroQ and placebo in individual domain scores from baseline at Day 60
The difference in change in brain-derived neurotrophic factor (BDNF) between NeuroQ and placebo | baseline (day 0) and 7 days
  The difference in change in brain-derived neurotrophic factor (BDNF) between NeuroQ and placebo from baseline at Day 7
The difference in change in BDNF between NeuroQ and placebo | baseline (day 0) and 60 days
  The difference in change in BDNF between NeuroQ and placebo from baseline at Day 60
The difference in change in C-reactive protein (CRP) between NeuroQ and placebo | baseline (day 0) and 60 days
  The difference in change in C-reactive protein (CRP) between NeuroQ and placebo from baseline at Day 60
The difference in change in memory between NeuroQ and placebo | baseline (day 0) and 60 days
  The difference in change in memory as assessed by the Everyday Memory Questionnaire questions 1, 2, and 18 between NeuroQ and placebo from baseline at Day 60

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events (AE) | baseline (day 0) and 60 days
  Incidence of pre-emergent and post-emergent adverse events (AE)
Clinically relevant changes in complete blood count after supplementation | baseline (day 0) and 60 days
  Clinically relevant changes in complete blood count after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in aspartate aminotransferase (AST) after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in alanine aminotransferase (ALT) after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in alkaline phosphatase (ALP) after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in total bilirubin after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in creatinine after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in sodium after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in potassium after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in chloride after supplementation
Clinically relevant changes in clinical chemistry | baseline (day 0) and 60 days
  Clinically relevant changes in estimated glomerular filtration rate (eGFR) after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No